CLINICAL TRIAL: NCT07286747
Title: A Phase II, Randomised, Double-blind, Placebo-controlled Trial to Evaluate the Efficacy and Safety of Oral Controlled-ileal-release Nicotinic Acid (CIR-NA) for Inducing Remission in Subjects With Prediabetes
Brief Title: Efficacy and Safety of Oral Controlled-release Nicotinic Acid (CIR-NA) for the Remission of Prediabetes. (CONCEPT)
Acronym: CONCEPT
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CONCEPT; LA1347/6-1 (Other Grant/Funding Number: German Research Foundation); 2024-519903-88-00 (EU CTIS Number)
Record Dates: First submitted 2025-12-03; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Prediabetes (Insulin Resistance, Impaired Glucose Tolerance)
MeSH Terms: conditions — Prediabetic State; Insulin Resistance; Glucose Intolerance

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CIR-NA 200 (Active Comparator): CIR-NA 200 mg once daily
  Interventions: Drug: controlled-ileal-release nicotinic acid as multiple dose 200 mg/day
- CIR-NA Placebo (Placebo Comparator): Placebo once daily
  Interventions: Drug: controlled-ileal-release nicotinic acid as multiple dose placebo
- CIR-NA 100 (Active Comparator): CIR-NA 100 mg once daily
  Interventions: Drug: controlled-ileal-release nicotinic acid as multiple dose 100 mg/day

INTERVENTIONS:
Drug: controlled-ileal-release nicotinic acid as multiple dose 100 mg/day — 130 participants will receive CIR-NA (100 mg/d). Additionally, all participants will receive standardized lifestyle recommendations regarding nutrition and physical activity.
  Other Names: CIR-NA 100 mg
  Arms: CIR-NA 100
Drug: controlled-ileal-release nicotinic acid as multiple dose 200 mg/day — 130 participants will receive CIR-NA (200 mg/d). Additionally, all participants will receive standardized lifestyle recommendations regarding nutrition and physical activity.
  Other Names: CIR-NA 200 mg
  Arms: CIR-NA 200
Drug: controlled-ileal-release nicotinic acid as multiple dose placebo — 130 participants will receive placebo. Additionally, all participants will receive standardized lifestyle recommendations regarding nutrition and physical activity.
  Other Names: Placebo
  Arms: CIR-NA Placebo

SUMMARY:
The goal of this clinical trial is to prevent the change from prediabetes (a pre-stage of type 2 diabetes mellitus (T2DM)) to T2DM in participants with prediabetes using oral CIR-NA (a nicotinic acid formulation that is designed to be released after reaching the ileum) which targeted the gut microbiota. The main questions it aims to answer are:

1. Is CIR-NA effective and does it prevent the change from prediabetes to T2DM?
2. Is the safety of CIR-NA that was observed in the Phase I clinical trial confirmed in subjects with prediabetes?

Researchers will compare CIR-NA to a placebo (a look-alike substance that contains no drug) in terms of an extended safety evaluation including safety laboratory assessments, physical examination, vital signs and 12-lead ECG.

Participants will:

Take CIR-NA or a placebo every day for 26-weeks. Visit the clinic at week 1 and subsequently once every 4 weeks for checkups and tests.

Receive standardized lifestyle recommendations regarding nutrition and physical activity during the intervention.

DETAILED DESCRIPTION:
The study is a multi-centre, randomised, double-blind, placebo-controlled trial evaluating the efficacy and safety of CIR-NA in participants with prediabetes. The trial includes a 26-week intervention period, which is expected to provide adequate time for prediabetes remission and a 4-week follow-up (FU) period.

A total of 390 male and female participants with a BMI of ≥ 20 kg/m² with prediabetes will be random-ised into three arms with 130 participants each in the CIR-NA (100 mg/d or 200 mg/d CIR-NA) and placebo groups. During the intervention, two indistinguishable tablets (CIR-NA and/or placebo) will be administered orally once daily. After screening and baseline assessment (including randomisation and IMP dispensing), 7 regular visits during treatment and one FU visit after 4 weeks are scheduled.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants ≥ 18 to < 80 years of age (at the time of signing the informed consent).
2. Body mass index ≥ 20 kg/m².
3. Ability to understand and comply with the protocol.
4. Signed written informed consent.
5. Diagnosed prediabetes according to the current EASD/DDG guidelines. Prediabetes is present if at least one value is in the prediabetes range, but no value is in the T2DM range.
6. Subgroup-specific: MASLD fibrosis score ≥ -1.455.

Exclusion Criteria:

1. Presence or a history of type 2 diabetes mellitus according to the current EASD/DDG guidelines.
2. Participants with relevant medical conditions (based on evaluation of medical history and screening assessments), unstable and uncontrolled underlying diseases, e.g., hypothyroidism, asthma, COPD or arterial hypertension, can be excluded per judgment of the Investigator.
3. Renal impairment (glomerular filtration rate <60 ml/min/1.73).
4. Impairment of hepatic function (one or more of liver enzymes alanine transaminase, aspartate transaminase and gamma glutamyl transferase [> 3-fold compared to normal range]).
5. Current infection with hepatitis B or C.
6. Clinically relevant abnormal findings in medical history or screening assessments which, in the opinion of the Investigator, may put the participant at risk when participating in the trial or provide difficulties in interpreting the trial data.
7. Current or history of malignancy except for completely resected basal cell carcinoma and squamous cell carcinoma of the skin.
8. Alcohol or drug abuse within the last 2 years at the discretion of the Investigator.
9. Subgroup-specific: Any circumstances which could contradict MRI and MRS imaging. For details, see Informed Consent Form (ICF) for additional examinations.
10. Regular use of any prescribed or over-the-counter medication, food supplements or herbal preparations, which cannot be terminated 3 weeks before baseline and during the full duration of the trial. Pain medication (e.g., ibuprofen or paracetamol), topical allergy medicines, hormone replacement therapies and oral contraceptives according to label are allowed. Medications in stable doses for controlling stable underlying diseases (see exclusion criterion 2) are also allowed per judgment of the Investigator.
11. Use of antibiotics (systemic or gut-acting [non-absorbed]) within 8 weeks prior to the first dose of IMP.
12. Long term use of higher doses of proton pump inhibitors, targeted H2-receptor antagonists or antacid formulations (i.e., doses equivalent to > 40 mg pantoprazole per day).
13. Known hypersensitivity towards any component of the CIR-NA or placebo tablets.
14. Participation in a clinical trial (as defined in the clinical trial regulation (CTR)), currently or within 4 weeks prior to screening for this trial or intake of an IMP within the last 8 weeks or 5 half-lives (whichever is longer) prior to screening (or longer, if necessary, at the Investigator's discretion).
15. Participants under legal supervision or guardianship, including participants who are committed to an institution by virtue of an order issued either by the judicial or the administrative authorities.
16. Participants who are dependent on the Investigator or the Sponsor.
17. Pregnant or breastfeeding women.
18. Women of childbearing potential (WoCBP) not using highly effective contraception till at least 1 month after last dosing of IMP.
19. Male participants with female partners of childbearing potential who are not willing to use a highly effective contraception till at least 1 month after last dosing of IMP.
20. Any other circumstances or medical conditions which could contradict a trial participation and lead the Investigator to assess the participant as unsuitable for trial participation.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-05-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Remission of prediabetes at week 26 | up to 185 days
  Remission of prediabetes at week 26 has been achieved when all values of HbA1c, fasting plasma glucose and 2-h-oGTT glucose are in the healthy range according to EASD/DDG guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Laudes, Prof. Dr., Principal Investigator — University Medical Center Schleswig-Holstein, Campus Kiel
Locations (1):
- University Medical Center Schleswig-Holstein, Campus Kiel, Kiel, Germany

IPD SHARING:
Plan to Share IPD: No